CLINICAL TRIAL: NCT02238457
Title: Effects of Low-Dose vs High-dose Losartan on Sympathetic Hyperactivity in Patients With Congestive Heart Failure
Brief Title: Study of High Dosage of Losartan in Comparison to Low Dose of Losartan in Heart Failure Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty recruiting patients
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Principal Investigator, Markus Schlaich, A/Prof, Baker Heart and Diabetes Institute
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Project 103-10
Record Dates: First submitted 2012-06-04; First posted 2014-09-12 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Heart Failure
Keywords: Heart failure; Losartan
MeSH Terms: conditions — Heart Failure | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose losartan (Active Comparator): Low dose losartan
  Interventions: Drug: Low dose losartan
- High dose losartan (Active Comparator): High dose losartan
  Interventions: Drug: High dose losartan

INTERVENTIONS:
Drug: Low dose losartan — 25 mg losartan bid for 10 weeks
  Other Names: losartan (Cozaar)
  Arms: Low dose losartan
Drug: High dose losartan — 50 mg, 75 mg, or 100 mg bid for 10 weeks. Dose will be determined by the medical doctor depending on patients' tolerability
  Other Names: Losartan (Cozaar)
  Arms: High dose losartan

SUMMARY:
The sympathetic nervous system, a part of the nervous system that stimulates the heart via release of substances, noradrenaline and adrenaline (combined called catecholamines), becomes activated in people with heart failure. As these people become sicker, the nervous system becomes more active, causing further damage to the heart.

Large trials have shown that Angiotensin-converting enzyme (ACE) inhibitors reduce morbidity and mortality in patients with heart failure. Higher doses of these drugs are more effective than lower doses. Studies show that ACE-inhibitors decrease catecholamine levels. This could be why congestive heart failure (CHF) patients taking this class of drugs show improvement in heart function.

There are several ways of measuring the activity of the sympathetic nervous system. The most common measurement is to test the blood for catecholamine levels. This is not very reliable or reproducible. Microneurography is a new technique used to measure sympathetic nerve activity. A small electrode (comparable to an acupuncture needle) is placed in a muscle nerve and hooked up to a stimulator and a recorder. It produces direct recordings of skeletal muscle nerve traffic. Both the rate and amplitude of the burst can be measured. The results in this technique are highly reproducible. By using this technique we get a more accurate picture of how the nervous system responds to medications given to treat heart failure.

Losartan (Cozaar) is an angiotensin II type 1 (AT1) receptor blocker. It blocks the binding of angiotensin II, a hormone that constricts blood vessels. As a result the blood vessels remain relaxed, leading to a reduction in the workload of the heart. Minor decreases in blood catecholamine levels have been reported with a low dose of this drug. The purpose of this study is to see whether a high dose of losartan (200 mg) has a greater effect on the sympathetic nervous system than a low dose of losartan (50 mg) does.

A total of 30 participants will be recruited. Participants will be assigned to one of two groups: high-dose, in which subjects will receive treatment of 200 mg/day of losartan, and low-dose, in which subjects will receive treatment of 50 mg/day of losartan. Via microneurography the investigators will measure the difference in sympathetic activity in subjects in high-dose vs low-dose losartan. The investigators expect to see further decrease in sympathetic activity in high-dose group than in low-dose group.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age between 21 and 75 years
* Diagnosis of mild to moderate congestive heart failure
* Coronary angiography identifying coronary artery disease as the likely cause of congestive heart failure
* Left Ventricular (LV) ejection fraction between 20 to 40 percent on echocardiography or RNA
* Sinus rhythm

Exclusion Criteria:

* Insulin-dependent diabetes mellitus
* Hypertension (higher than 140/90 mmHg at rest)
* Use of sympatholytic agents such as clonidine, methyldopa, reserpine
* Significant non-cardiac disease, possibly affecting cardiovascular regulation
* Autonomic neuropathy of any cause
* Leg injuries with nerve damage
* Poor bladder control
* Recent history of alcoholism, drug abuse, significant psychiatric disorders
* Known adverse events to AT1-receptor blockers
* Unlikely to tolerate being off digoxin and off blockers of the RAS for a short period
* Ischemic event within past 3 months
* Serum creatinine higher than 200 mmol/L
* Patients taking digoxin for atrial fibrillation
* Patients who require treatment with aldactone
* Patients with more than mild stable angina while on beta-blockers and/or calcium antagonists
* Patients on coumadin

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Effect of losartan on the sympathetic nervous system. | 10 weeks
  Assessed by microneurographic recordings of muscle sympathetic nerve activity from the peroneal nerve.

SECONDARY OUTCOMES:
Change in plasma catecholamines. | 10 weeks
  Plasma catecholamines will be measured by High-performance liquid chromatography (HPLC). Samples will be collected for plasma aldosterone, plasma renin and plasma angiotensin II.
Change in central hemodynamics. | 10 weeks
  Invasive measurement of central hemodynamic parameters; heart rate, blood pressure, cardiac output (CO), pulmonary capillary wedge pressure (PCWP), right arterial pressure (RAP).

CONTACTS AND LOCATIONS:
Overall Officials: Markus P Schlaich, Principal Investigator — Baker IDI Heart & Diabetes Institute